CLINICAL TRIAL: NCT03332511
Title: A Phase 4 Study of Nilotinib in Korean Patients With Philadelphia Chromosome-positive Chronic Myeloid Leukemia in Chronic Phase
Brief Title: Efficacy and Safety of Nilotinib in CML-CP
Acronym: ENESTKorea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Inho Kim, Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1110-124-383
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational arm (Experimental): Oral nilotinib 300mg twice daily with a 12-hour interval
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Nilotinib 300mg twice-daily
  Other Names: Tasigna

SUMMARY:
ENESTKorea is a phase 4, multi-institutional, single-arm, open-label study investigating the efficacy and safety of nilotinib at the currently approved dose (300 mg twice daily) and its exposure-outcome relationship, in adult patients diagnosed as Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase.

DETAILED DESCRIPTION:
Nilotinib is a second-generation tyrosine kinase inhibitor with improved efficacy compared to imatinib. However, there are still many patients for whom the therapeutic response is inadequate, or toxicity is limiting the treatment. Serum concentration of nilotinib was shown to affect time to response and progression in previous studies. Therefore, the investigators hypothesized that the optimal plasma level of nilotinib that is sufficient to achieve adequate clinical response while not generating major adverse events could be elucidated by the analysis of combined clinical and pharmacokinetic data.

ENESTKorea is a phase 4, multi-institutional, single-arm, open-label study investigating the efficacy and safety of nilotinib at the currently approved dose (300 mg twice daily), in adult patients diagnosed as Philadelphia chromosome (Ph)-positive chronic myeloid leukemia in chronic phase (CML-CP). Plasma samples are collected every three months, for up to 12 months, to determine plasma nilotinib concentrations (PNCs). The primary endpoint is the cumulative rate of molecular response 4.5 (MR4.5; BCR-ABL1IS ≤ 0.0032%) by 24 months. Secondary endpoints include the cumulative rates of MR3 (BCR-ABLIS ≤ 0.1%) and MR4 (BCR-ABLIS ≤ 0.01%) by 12 and 24 months; time to MR3, MR4, and MR4.5; progression-free survival (PFS); overall survival (OS). Correlations between PNCs and clinical outcomes are also analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Aged 19 or older
* Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase

Exclusion Criteria:

* CML with atypical BCR-ABL1 transcripts (transcripts other than e13a2 or e14a2)
* Eastern Cooperative Oncology Group performance status ≥ 3
* Cardiac abnormality including a corrected QT interval ≥ 480 milliseconds, complete left bundle branch block, permanent pacemaker implantation, congenital long QT syndrome, history of tachyarrhythmia requiring treatment, clinically significant resting bradycardia, history of acute coronary syndrome within 12 months, and decompensated congestive heart failure
* Organ dysfunction defined by total serum bilirubin levels ≥ 1.5 × the upper limit of the normal range (ULN), creatinine ≥ 1.5 × ULN, aspartate or alanine aminotransferase ≥ 2.5 × ULN, amylase or lipase ≥ 1.5 × ULN and alkaline phosphatase ≥ 2.5 × ULN not directly related to the CML
* Uncontrolled hypertension and/or diabetes
* Active and uncontrolled infection
* Major surgery within two weeks or incomplete recovery from the previous surgery
* Congenital or acquired bleeding tendency
* Impaired gastrointestinal absorption
* History of small bowel resection or bypass surgery
* History of acute pancreatitis within 12 months or chronic pancreatitis
* Concomitant administration of strong irreplaceable CYP3A4 inhibitors or inducers, QT-prolonging agents, or coumarin derivatives
* Any other uncontrolled medical conditions that would present substantial safety risks or compromise compliance with the study treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

PRIMARY OUTCOMES:
Cumulative rate of molecular response 4.5 by 24 months | 24 months
  Cumulative rate of BCR-ABL1 fusion transcripts ≤ 0.0032%, measured by real-time quantitative polymerase chain reaction and standardized to the international scale

SECONDARY OUTCOMES:
Cumulative rate of molecular response 3 by 24 months | 24 months
  Cumulative rate of BCR-ABL1 fusion transcripts ≤ 0.1%, measured by real-time quantitative polymerase chain reaction and standardized to the international scale
Cumulative rate of molecular response 3 by 12 months | 12 months
  Cumulative rate of BCR-ABL1 fusion transcripts ≤ 0.1%, measured by real-time quantitative polymerase chain reaction and standardized to the international scale
Cumulative rate of molecular response 4 by 24 months | 24 months
  Cumulative rate of BCR-ABL1 fusion transcripts ≤ 0.01%, measured by real-time quantitative polymerase chain reaction and standardized to the international scale
Cumulative rate of molecular response 4 by 12 months | 12 months
  Cumulative rate of BCR-ABL1 fusion transcripts ≤ 0.01%, measured by real-time quantitative polymerase chain reaction and standardized to the international scale
Progression-free survival | 24 months
  Time from enrollment to documented disease progression or death from any cause
Overall survival | 24 months
  Time from enrollment to death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Inho Kim, MD, Principal Investigator — Seoul National University Hospital

IPD SHARING:
Plan to Share IPD: No
Individual participant data are not currently planned to be shared.

REFERENCES:
- [Derived] Shin J, Koh Y, Yoon SH, Cho JY, Kim DY, Lee KH, Kim HJ, Ahn JS, Kim YK, Park J, Sohn SK, Moon JH, Lee YJ, Yoon S, Lee JO, Cheong JW, Kim KH, Kim SH, Kim HG, Kim H, Nam SH, Do YR, Park SG, Park SK, Bae SH, Song HH, Shin DY, Oh D, Kim MK, Jung CW, Park S, Kim I. A phase 4 study of nilotinib in Korean patients with Philadelphia chromosome-positive chronic myeloid leukemia in chronic phase: ENESTKorea. Cancer Med. 2018 May;7(5):1814-1823. doi: 10.1002/cam4.1450. Epub 2018 Mar 25. PMID 29577674